CLINICAL TRIAL: NCT01238575
Title: Guanfacine for the Treatment of Hyperactivity in Pervasive Developmental Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Emory University (Other); Massachusetts General Hospital (Other); Seattle Children's Hospital (Other); University of California, Los Angeles (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1001006172; R01MH083707 (NIH)
Record Dates: First submitted 2010-10-29; First posted 2010-11-10 (Estimated); Results first posted 2015-12-07 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Pervasive Development Disorders
Keywords: Pervasive Developmental Disorders; PDD; PDD-NOS; Autistic Disorder; Autism; Asperger's Disorder; Hyperactivity; Attention Deficit Hyperactivity Disorder; ADHD; Medication; Drug; Guanfacine; Intuniv; Placebo; Methylphenidate
MeSH Terms: conditions — Child Development Disorders, Pervasive; Autistic Disorder; Asperger Syndrome; Spasm; Attention Deficit Disorder with Hyperactivity | interventions — Guanfacine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Extended-release guanfacine (Experimental)
  Interventions: Drug: extended-release guanfacine
- Inactive placebo (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Other: placebo — Administered for up to 8 weeks.
  Arms: Inactive placebo
Drug: extended-release guanfacine — 1 mg tablets; flexible dosing up to 4 mg/day for up to 16 weeks
  Other Names: Intuniv
  Arms: Extended-release guanfacine

SUMMARY:
The purpose of this study is to determine whether guanfacine (trade name Intuniv) by itself or in combination with methylphenidate (also known as Ritalin) is helpful for treating hyperactivity in children and adolescents with a Pervasive Developmental Disorders (PDDs).

DETAILED DESCRIPTION:
Pervasive Developmental Disorders (PDDs) are a group of conditions that includes Autistic Disorder, Asperger's disorder and so called Pervasive Developmental Disorder - Not Otherwise Specified. Children with PDD show delays in speech and language and reduced social interaction. Some children with PDD have also have problems with overactivity, impulsiveness and distractability. These behaviors are seen in children with Attention Deficit Hyperactivity Disorder (ADHD). Extended release guanfacine (Intuniv) is FDA-approved for the treatment of children with ADHD. The purpose of this study is to evaluate whether Intuniv is an effective treatment for ADHD symptoms in children with PDD.

This study has four parts: an 8-week double-blind trial, an 8-week blinded extension phase (for positive responders only), an 8-week open-label trial, and a 4-week add-on study. Following confirmation of eligibility, participants will be randomly assigned to receive either guanfacine or placebo in the 8-week double-blind trial. Children who show improvement after 8 weeks of treatment will continue on their assigned treatment for an additional 8 weeks (blinded extension phase). Children who show partial improvement with guanfacine will be offered 4 weeks of treatment with guanfacine plus methylphenidate (add-on study). Children who show no improvement on placebo will be offered 8 weeks of treatment with guanfacine (open-label trial). Children who show no improvement on guanfacine will exit the study.

Side effects and treatment response will be assessed at regularly scheduled visits.

The study protocol was formally revised with the Yale University IRB in May 2013 to address an early close to enrollment due to a reduction in funding. The original anticipated enrollment numbers of 112 subjects was reduced to 60 subjects. The study statistician was consulted prior to enrollment closure to address any issues related to statistical power and the adjustments made to the final statiscal analysis plan.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PDD (PDD-NOS, Asperger's Disorder, Autistic Disorder)
* Hyperactivity
* Between ages 5 years 0 months and 13 years 11 months.
* Weight >/= 15 kg (33 lb)
* A mental age of at least 18 months

Exclusion Criteria:

* Prior failed treatment with an adequate trial of guanfacine in the last 2 years
* Concurrent treatment with another psychoactive medication

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2011-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Scahill, MSN, PhD, Principal Investigator — Emory University; James McCracken, MD, Principal Investigator — University of California, Los Angeles; Bryan King, MD, Principal Investigator — Seattle Children's Hospital; Christopher McDougle, MD, Principal Investigator — Massachusetts General Hospital; James Dziura, MPH, PhD, Principal Investigator — Yale University
Locations (5):
- United States (5):
  - University of California, Los Angeles, Los Angeles, California
  - Yale University, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - Massachusetts General Hospital, Lexington, Massachusetts
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- [Background] Scahill L, Aman MG, McDougle CJ, McCracken JT, Tierney E, Dziura J, Arnold LE, Posey D, Young C, Shah B, Ghuman J, Ritz L, Vitiello B. A prospective open trial of guanfacine in children with pervasive developmental disorders. J Child Adolesc Psychopharmacol. 2006 Oct;16(5):589-98. doi: 10.1089/cap.2006.16.589. PMID 17069547
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 81 total patients screened. 13 ineligible. 6 Declined
Period: Overall Study
Arm/Group | Extended-release Guanfacine | Inactive Placebo
Started | 30 | 32
Completed | 26 | 28
Not Completed | 4 | 4
Not completed — Lack of Efficacy | 2 | 4
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Extended-release Guanfacine | Inactive Placebo | Total
Number analyzed (Participants) | 30 | 32 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.44 (2.28) | 8.39 (2.23) | 8.4 (2.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 26 | 27 | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 7 | 4 | 11
  White | 17 | 23 | 40
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Aberrant Behavior Checklist Hyperactivity Subscale
Description: The Aberrant Behavior Checklist (ABC) is a symptom checklist for assessing problem behaviors in individuals ages 6 to 54 with mental retardation. The full ABC is a 58-item parent-rating with five factors: Irritability, Social Withdrawal, Stereotypy, Hyperactivity and Inappropriate Speech. The 16-item Hyperactivity subscale covers over-activity (7 items), impulsiveness (2 items), inattention (3 items) and noncompliance (4 items). It has been used as a primary outcome measure in several trials of children with developmental disabilities. The interpretation of the tool and its sub-scales is that a greater number of items, indicates greater severity. The range of scores is 0 to 48.
Time Frame: Week 8
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Extended-release Guanfacine | Inactive Placebo
Number analyzed (Participants) | 30 | 32
units on a scale | 19.3 [15.33 to 23.33] | 29.7 [25.82 to 33.53]

2. Secondary Outcome: ADHD Rating Scale - Total
Description: The ADHD Rating Scale (ADHD-RS) is an 18-item scale directly derived from DSM-IV criteria for Attention Deficit Hyperactivity Disorder with established reliability, validity and sensitivity to change. The ADHD Rating Scale-IV is completed independently by the parent and scored by a clinician. The scale consists of 2 subscales: inattention (9 items) and hyperactivity-impulsivity (9 items). If 3 or more items are skipped, the clinician should use extreme caution in interpreting the scale. Results from this rating scale alone should not be used to make a diagnosis. The total score can range from 0 to 54, with a higher score indicating greater severity.
Time Frame: Week 8
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Extended-release Guanfacine | Inactive Placebo
Number analyzed (Participants) | 30 | 32
units on a scale | 25.2 [21.44 to 29.03] | 38.0 [34.44 to 41.63]

3. Secondary Outcome: Aberrant Behavior Checklist Irritability Subscale
Description: The Aberrant Behavior Checklist (ABC) is a symptom checklist for assessing problem behaviors in individuals ages 6 to 54 with mental retardation. It is a 58 item checklist which takes about 10 - 15 minutes to complete. There are five subscales: a) Irritability and Agitation b) Lethargy and Social Withdrawal c) Stereotypic Behavior d) Hyperactivity and Noncompliance and e) Inappropriate Speech. The higher the number of items (score), the greater the amount of symptoms. Scores can range from 0 to 45.
Time Frame: 8 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Extended-release Guanfacine | Inactive Placebo
Number analyzed (Participants) | 30 | 32
units on a scale | 13.5 [10.01 to 17.06] | 16.1 [12.68 to 19.54]

4. Secondary Outcome: Aberrant Behavior Checklist Social Withdrawal Subscale
Description: The Aberrant Behavior Checklist (ABC) is a symptom checklist for assessing problem behaviors in individuals ages 6 to 54 with mental retardation. The full ABC is a 58-item parent-rating with five factors: Irritability, Social Withdrawal, Stereotypy, Hyperactivity and Inappropriate Speech. It has been used as a primary outcome measure in several trials of children with developmental disabilities. The interpretation of the tool and its sub-scales is that a greater number of items, indicates greater severity. This subscale's scores can range from 0 to 48.
Time Frame: 8 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Extended-release Guanfacine | Inactive Placebo
Number analyzed (Participants) | 30 | 32
units on a scale | 9.8 [7.26 to 12.27] | 8.6 [6.10 to 11.02]

5. Secondary Outcome: Aberrant Behavior Checklist Sterotypy Subscale
Description: The Aberrant Behavior Checklist (ABC) is a symptom checklist for assessing problem behaviors in individuals ages 6 to 54 with mental retardation. The full ABC is a 58-item parent-rating with five factors: Irritability, Social Withdrawal, Stereotypy, Hyperactivity and Inappropriate Speech. It has been used as a primary outcome measure in several trials of children with developmental disabilities. The interpretation of the tool and its sub-scales is that a greater number of items, indicates greater severity. This subscale's scores can range from 0 to 21.
Time Frame: 8 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Extended-release Guanfacine | Inactive Placebo
Number analyzed (Participants) | 30 | 32
units on a scale | 3.6 [2.03 to 5.26] | 5.9 [4.37 to 7.49]

6. Secondary Outcome: Aberrant Behavior Checklist Inappropriate Speech Subscale
Description: The Aberrant Behavior Checklist (ABC) is a symptom checklist for assessing problem behaviors in individuals ages 6 to 54 with mental retardation. The full ABC is a 58-item parent-rating with five factors: Irritability, Social Withdrawal, Stereotypy, Hyperactivity and Inappropriate Speech. It has been used as a primary outcome measure in several trials of children with developmental disabilities. The interpretation of the tool and its sub-scales is that a greater number of items, indicates greater severity. This subscale's scores can range from 0 to 12.
Time Frame: 8 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Extended-release Guanfacine | Inactive Placebo
Number analyzed (Participants) | 30 | 32
units on a scale | 4.2 [3.24 to 5.26] | 5.99 [4.5 to 6.97]

7. Secondary Outcome: ADHD Rating Scale - Inattention Subscale
Description: The ADHD Rating Scale (ADHD-RS) is an 18-item scale directly derived from DSM-IV criteria for Attention Deficit Hyperactivity Disorder with established reliability, validity and sensitivity to change. The ADHD Rating Scale-IV is completed independently by the parent and scored by a clinician. The scale consists of 2 subscales: inattention (9 items) and hyperactivity-impulsivity (9 items). If 3 or more items are skipped, the clinician should use extreme caution in interpreting the scale. Results from this rating scale alone should not be used to make a diagnosis. This subscale can range from 0 to 27 for scoring, with a higher score indicating greater severity.
Time Frame: 8 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Extended-release Guanfacine | Inactive Placebo
Number analyzed (Participants) | 30 | 32
units on a scale | 14.7 [12.55 to 16.78] | 19.5 [17.52 to 21.56]

8. Secondary Outcome: ADHD Rating Scale - Hyperactivity Subscale
Description: The ADHD Rating Scale (ADHD-RS) is an 18-item scale directly derived from DSM-IV criteria for Attention Deficit Hyperactivity Disorder with established reliability, validity and sensitivity to change. The ADHD Rating Scale-IV is completed independently by the parent and scored by a clinician. The scale consists of 2 subscales: inattention (9 items) and hyperactivity-impulsivity (9 items). If 3 or more items are skipped, the clinician should use extreme caution in interpreting the scale. Results from this rating scale alone should not be used to make a diagnosis. This subscale can range from 0 to 27 for scoring,with a higher score indicating greater severity.
Time Frame: 8 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Extended-release Guanfacine | Inactive Placebo
Number analyzed (Participants) | 30 | 32
units on a scale | 10.6 [8.5 to 12.75] | 18.7 [16.66 to 20.69]

9. Secondary Outcome: Aberrant Behavior Checklist Hyperactivity Subscale
Description: as for outcome 1
Time Frame: Baseline
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Extended-release Guanfacine | Inactive Placebo
Number analyzed (Participants) | 30 | 32
units on a scale | 34.4 [32.4 to 36.4] | 34.25 [31.74 to 36.76]

10. Secondary Outcome: Aberrant Behavior Checklist Irritability Subscale
Description: The Aberrant Behavior Checklist (ABC) is a symptom checklist for assessing problem behaviors in individuals ages 6 to 54 with mental retardation. The full ABC is a 58-item parent-rating with five factors: Irritability, Social Withdrawal, Stereotypy, Hyperactivity and Inappropriate Speech. It has been used as a primary outcome measure in several trials of children with developmental disabilities. The interpretation of the tool and its sub-scales is that a greater number of items, indicates greater severity. Scores for this subscale can range from 0 to 45.
Time Frame: Baseline
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Extended-release Guanfacine | Inactive Placebo
Number analyzed (Participants) | 30 | 32
units on a scale | 20.3 [16.79 to 23.81] | 18.06 [14.54 to 21.58]

11. Secondary Outcome: Aberrant Behavior Checklist Social Withdrawal Subscale
Description: as for outcome 4
Time Frame: Baseline
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Extended-release Guanfacine | Inactive Placebo
Number analyzed (Participants) | 30 | 32
units on a scale | 13.6 [10.08 to 17.12] | 12.06 [8.71 to 15.41]

12. Secondary Outcome: Aberrant Behavior Checklist Sterotypy Subscale
Description: as for outcome 5
Time Frame: Baseline
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Extended-release Guanfacine | Inactive Placebo
Number analyzed (Participants) | 30 | 32
units on a scale | 8.53 [6.41 to 10.66] | 9.31 [7.31 to 11.32]

13. Secondary Outcome: Aberrant Behavior Checklist Inappropriate Speech Subscale
Description: as for outcome 6
Time Frame: Baseline
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Extended-release Guanfacine | Inactive Placebo
Number analyzed (Participants) | 30 | 32
units on a scale | 6.33 [5.02 to 7.65] | 6.84 [5.63 to 8.06]

14. Secondary Outcome: ADHD Rating Scale - Inattention Subscale
Description: as for outcome 7
Time Frame: Baseline
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Extended-release Guanfacine | Inactive Placebo
Number analyzed (Participants) | 30 | 32
units on a scale | 20.53 [19.17 to 21.9] | 20.41 [18.75 to 22.06]

15. Secondary Outcome: ADHD Rating Scale - Hyperactivity Subscale
Description: as for outcome 7
Time Frame: Baseline
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Extended-release Guanfacine | Inactive Placebo
Number analyzed (Participants) | 30 | 32
units on a scale | 19.00 [17.38 to 20.62] | 19.5 [17.71 to 21.29]

16. Secondary Outcome: ADHD Rating Scale - Total
Description: as for outcome 2
Time Frame: Baseline
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Extended-release Guanfacine | Inactive Placebo
Number analyzed (Participants) | 30 | 32
units on a scale | 39.53 [37.33 to 41.73] | 39.91 [37.5 to 42.32]

ADVERSE EVENTS:
Arm/Group | Extended-release Guanfacine | Inactive Placebo
Serious Adverse Events (participants affected / at risk) | 1/30 | 0/32
Other Adverse Events (participants affected / at risk) | 30/30 | 25/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Extended-release Guanfacine (N=30) | Inactive Placebo (N=32)
Aggressive (Psychiatric disorders) | 1 | 0 — Subject became verbally and physically agressive
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Extended-release Guanfacine (N=30) | Inactive Placebo (N=32)
Drowsiness (Nervous system disorders) | 26 | 3
Fatigue (General disorders) | 19 | 3
Decreased Appetite (General disorders) | 13 | 2
Emotional/tearful (General disorders) | 12 | 3
Dry Mouth (Gastrointestinal disorders) | 12 | 1
Irritability (General disorders) | 11 | 3
Anxiety (Psychiatric disorders) | 9 | 1
Headache (Nervous system disorders) | 9 | 6
Increased Energy (General disorders) | 9 | 6
Mid sleep awakening (Psychiatric disorders) | 9 | 2
Stomachache (Gastrointestinal disorders) | 8 | 4
Constipation (Gastrointestinal disorders) | 7 | 2
Increased Repetitive Behavior (Psychiatric disorders) | 5 | 3
Aggression (Psychiatric disorders) | 5 | 2
Depressed Mood (Psychiatric disorders) | 4 | 1
Cough/Congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Self-injury (Psychiatric disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 3 | 2
Trouble Falling Asleep (Psychiatric disorders) | 3 | 2
Dizziness (Nervous system disorders) | 3 | 2
Silly (Psychiatric disorders) | 3 | 5
Weakness (General disorders) | 3 | 1
Diarrhea (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 3 | 3
Increased Appetite (Gastrointestinal disorders) | 2 | 2
Excessive Talking (Psychiatric disorders) | 2 | 9
Blurred Vision (Eye disorders) | 2 | 0
Skin rash/Eczema (Skin and subcutaneous tissue disorders) | 2 | 4
Nightmares (Psychiatric disorders) | 2 | 0
Enuresis (Renal and urinary disorders) | 2 | 2
Motor Tics (Nervous system disorders) | 1 | 2
Skin Picking (Skin and subcutaneous tissue disorders) | 1 | 3
Fever (General disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No